CLINICAL TRIAL: NCT06190665
Title: DEB-TACE With Visualable Microspheres Versus PVA Microspheres for Hepatocellular Carcinoma: a Prospective, Multicenter, Randomized Controlled, Non-inferior Trial
Brief Title: DEB-TACE With Visualable Microspheres Versus PVA Microspheres for HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dean, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHANCE 2305
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; TACE; Microspheres
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: DEB-TACE with visualable microspheres or PVA microspheres
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visualable microspheres (Experimental): DEB-TACE with visualable microspheres
  Interventions: Device: DEB-TACE with visualable microspheres
- PVA microspheres (Active Comparator): DEB-TACE with polyvinyl alcohol microspheres
  Interventions: Device: DEB-TACE with PVA microspheres

INTERVENTIONS:
Device: DEB-TACE with visualable microspheres — Drug-eluting Beads Transcatheter Arterial Chemoembolization(DEB-TACE) with visualable microspheres
  Arms: Visualable microspheres
Device: DEB-TACE with PVA microspheres — Drug-eluting Beads Transcatheter Arterial Chemoembolization(DEB-TACE) with polyvinyl alcohol microspheres
  Arms: PVA microspheres

SUMMARY:
This study will evaluate the safety and efficacy of DEB-TACE with visualable embolization microspheres versus PVA microspheres for hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled, non-inferior trial to evaluate the safety and efficacy of DEB-TACE with visualable microspheres or PVA microspheres for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* CNLC Ia-IIIa HCC patients who require transarterial chemoembolization (TACE) and are not suitable for or refuse surgical resection, liver transplantation, or ablation Liver function classification of Child-Pugh A or B
* ECOG PS score of 0-2
* With measurable lesions that had not been embolized (if there are more than 3 lesions, select the three largest lesions as target lesions, and the maximum diameter of target lesion is ≤10cm)
* Agree to participate in this trial and voluntarily sign the informed consent form

Exclusion Criteria:

* Target lesions were embolized, or will require concomitant ablation or radiotherapy after TACE treatment(s)
* With diffuse liver tumor or extrahepatic metastasis, expected survival <6 months With sepsis or multiple organ dysfunction
* Severe liver dysfunction (Child-Pugh C) , or severerenal dysfunction (blood creatinine >2 mg/dL)
* Significant reductions in white blood cells or platelets (white blood cells <3.0×10^9/L, platelets <50×10^9/L, hemoglobin<60g/L) that cannot be corrected (except splenomegaly or chemotherapy-induced bone marrow suppression) Uncorrectable coagulation dysfunction (PT prolonged by >3 seconds above the upper limit of normal)
* With severe infection (>5 times the upper limit of normal white blood cells) The main portal vein was completely embolized by tumor thrombus without collateral blood supply
* With risk of ectopic embolization (uncorrected arteriovenous fistula or portal venous fistula) in the target lesion supplying arteries
* Angiography shows vascular anatomy obstruction or vasospasm that will affect the catheter placemenr embolic agent injection
* Known allergy to iodine-containing contrast agents, polyvinyl alcohol materials or anthracycline t ochemotherapy drugs
* Pregnant or lactating women
* Patients who are participating in other trial(s)
* Unsuitable for participation in this trial deemed by the researchers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) for target lesions 1 month after the last TACE treatment | 1 month after last TACE treatment
  Target lesions were evaluated according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.

SECONDARY OUTCOMES:
Visualization score of embolic area | Immediately, 1 day, 1 month after first TACE treatment, and 1 month, 3 months, or 6 months since the last TACE treatment
  Evaluation will be performed, based on CBCT images after the first TACE treatment, or CT plain images after the last TACE treatment as follow: 3 points: dense imaging (imaging area >75% of tumor area); 2 points: mixed imaging (imaging area 25%-75% of tumor area); 1 point: weak imaging (imaging area <25% of tumor area); 0 point: not visible (no imaging in the tumor area).
Embolization success rate of target lesions | Immediately after each TACE treatment
  Defined as the number of successful embolizations for the target lesions / the total number of participants ×100%.
Equipment performance evaluation | From the begin to immediately after each TACE treatment
  Includes,the visualization performance of the microspheres on the fluoroscopy or cone-beam CT imaging; whether the microspheres can be easy pushed and pass through the catheter smoothly; whether the micro-catheter will be blocked during the process of pushing and releasing?
Disease control rate (DCR) for target lesions | 1 month after the first TACE treatment, and 3 months after the last TACE treatment
  Target lesions will be evaluated according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST), based on the enhanced CT/MRI (liver) images.
Objective response rate（ORR） | 1 month after the first TACE treatment and 1 month, 3 months since the last TACE treatment
  Target lesions will be evaluated according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST), based on the enhanced CT/MRI (liver) images.
Number of TACE treatments for target lesions | 6 month since the last TACE treatment
  Totel times of TACE treatments for all target lesions

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, Principal Investigator — Zhongda Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Zhongda Hospital，Southeast University, Nanjing, Jiangsu